CLINICAL TRIAL: NCT01410773
Title: Ninja 2 User Performance Evaluation
Brief Title: User Performance Evaluation of an Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R&D-2010-2011.32
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the System (Experimental): Untrained subjects with diabetes (at least 70% of subjects will be insulin users) use an investigational blood glucose monitoring system (Ninja 2) to self-test capillary blood obtained from fingerstick and palm.
  Interventions: Device: Ninja 2 Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: Ninja 2 Investigational Blood Glucose Monitoring System — The Ninja 2 meter is a Bayer investigational meter that uses an investigational sensor.

SUMMARY:
The purpose of this study is to demonstrate that untrained subjects with diabetes can use an investigational Blood Glucose Monitoring System (BGMS) with capillary blood obtained from fingerstick and from Alternative Site (AST) Palm .

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and above
* Diagnosed as having type 1 or type 2 diabetes
* Currently self-testing blood glucose at home
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Blood Borne infections like hepatitis or HIV or infections such as tuberculosis
* Hemophilia or any other bleeding disorder
* Employee of competitive medical device company,immediate family member of such, or living within the household of such
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simmons, MD, Principal Investigator — Ascensia Diabetes Care
Locations (1):
- Bayer HealthCare LLC, Diabetes Care, Mishawaka, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the System: Untrained subjects with diabetes (at least 70% of subjects will be insulin users) use an investigational blood glucose monitoring system (Ninja 2) to self-test capillary blood obtained from fingerstick and palm.
  Ninja 2 Investigational Blood Glucose Monitoring System : The Ninja 2 meter is a Bayer investigational meter that uses an investigational sensor.
Period: Overall Study
Arm/Group | Intended Users of the System
Started | 110
Completed | 110
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 110
Age, Customized [Mean (Full Range); unit: years]
  Mean (Full range of ages) | 53.1 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 52
Region of Enrollment [Number; unit: participants]
  United States | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG) Results Within +/-15mg/dL(<75 mg/dL) or Within +/- 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test fingerstick blood using an investigational Blood Glucose Meter (BGM). BGM results are compared with capillary plasma BG results obtained with a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG meter results are used to calculate the number of BG results within +/- 15mg/dL (for reference BG results <75mg/dL) or within +/- 20%(for reference BG results >=75mg/dL) of the reference method results (YSI capillary plasma).
Time Frame: 1 hour
Population: 110 subjects tested one of 3 test strip lots on the BGM system. 110 (1x110) test results are available.
Measure: Number; unit: participants
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 110
participants
  # within +/-15mg/dL(<75mg/dL)or 20% (>=75mg/dL) | 110
  # within +/-15mg/dL(<75mg/dL)or 15% (>=75mg/dL) | 109
  # within +/-10mg/dL(<75mg/dL)or 10% (>=75mg/dL) | 109
  # within +/-5mg/dL(<75mg/dL) or 5% (>=75mg/dL) | 90

2. Secondary Outcome: Number of Alternative Site (AST) Palm Blood Glucose (BG) Results Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test subject Alternative Site (AST) Palm blood using an investigational Blood Glucose Monitoring System (BGMS). BGM meter results are compared with capillary plasma BG results obtained with a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG meter results are used to calculate the number of BG results within +/- 15mg/dL (for reference BG results <75mg/dL) or +/- 20% (for reference BG results >=75mg/dL) of the YSI capillary plasma reference method results.
Time Frame: 1 hour
Population: One subject had low blood sugar. The protocol (and User Guide) do not allow alternative site testing when blood sugar is low. The remaining 109 subjects tested one strip lot on the BGM system. 109 test results were available.
Measure: Number; unit: participants
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 109
participants
  # within +/- 15mg/dL(<75mg/dL) or 20% (>=75mg/dL) | 106
  # within +/- 15mg/dL(<75mg/dL) or 15% (>=75mg/dL) | 105
  # within +/- 10mg/dL(<75mg/dL) or 10% (>=75mg/dL) | 97
  # within +/- 5mg/dL(<75mg/dL) or 5% (>=75mg/dL) | 67

ADVERSE EVENTS:
Time Frame: Each subject participated for approximately 1 hour.
Arm/Group | Intended Users of the System
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes